CLINICAL TRIAL: NCT01773408
Title: A Multi-Center, Open-Label, Phase 1/1b Study of Escalating Doses of RO5503781 Administered Orally as 1) a Single Agent, 2) In Combination With Cytarabine, or 3) With Cytarabine and Anthracycline and 4) Assessing PK and Safety of New Optimized Formulation of RO5503781 With Cytarabine in Patients With Acute Myelogenous Leukemia (AML)
Brief Title: A Study of RO5503781 as a Single Agent or in Combination With Cytarabine in Participants With Acute Myelogenous Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NP28679; 2012-004882-41 (EudraCT Number)
Record Dates: First submitted 2013-01-18; First posted 2013-01-23 (Estimated); Last update posted 2017-01-25 (Estimated); Status verified 2017-01

CONDITIONS: Myelogenous Leukemia, Acute
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Idarubicin; Daunorubicin; Cytarabine

ARMS (4):
- Part 1: RO5503781 (Experimental): Participants will receive RO5503781 alone in escalating doses on Days 1 to 5 of each 28-day cycle until disease progression or unacceptable toxicity.
  Interventions: Drug: RO5503781 MBP
- Part 2: RO5503781 + Cytarabine (Experimental): Participants will receive RO5503781 in escalating doses on Days 1 to 5 and cytarabine on Days 1 to 6 of each 28-day cycle until disease progression or unacceptable toxicity.
  Interventions: Drug: RO5503781 MBP; Drug: Cytarabine
- Part3:RO5503781+Cytarabine+Anthracycline (Experimental): Participants will receive RO5503781 on Days 1 to 5, cytarabine on Days 1 to 7, and anthracycline (daunorubicin or idarubicin) on Days 1 to 3 of each 28-day cycle until disease progression or unacceptable toxicity.
  Interventions: Drug: RO5503781 MBP; Drug: Idarubicin; Drug: Daunorubicin; Drug: Cytarabine
- Part 4: Optimized RO5503781 + Cytarabine (Experimental): Participants will receive optimized RO5503781 formulation on Days 1 to 5 and cytarabine on Days 1 to 6 of each 28-day cycle until disease progression or unacceptable toxicity.
  Interventions: Drug: RO5503781 SDP; Drug: Cytarabine

INTERVENTIONS:
Drug: RO5503781 MBP — Participants will receive RO5503781 tablets daily (current formulation) containing microprecipitated bulk powder (MBP) at a starting dose of 400 milligrams (mg).
  Arms: Part 1: RO5503781; Part 2: RO5503781 + Cytarabine; Part3:RO5503781+Cytarabine+Anthracycline
Drug: RO5503781 SDP — Participants will receive RO5503781 tablets daily (new optimized formulation) containing spray-dried powder (SDP) at recommended dose(s) for development from Phase 1b to Phase 3.
  Arms: Part 4: Optimized RO5503781 + Cytarabine
Drug: Idarubicin — Idarubicin will be administered as per standard clinical practice.
  Arms: Part3:RO5503781+Cytarabine+Anthracycline
Drug: Daunorubicin — Daunorubicin will be administered as per standard clinical practice.
  Arms: Part3:RO5503781+Cytarabine+Anthracycline
Drug: Cytarabine — Parts 2 and 4: Participants will receive cytarabine 1000 milligrams per meter squared (mg/m^2) intravenous (IV) infusion daily. Part 3: Participants will receive cytarabine 100-200 mg/m^2 IV infusion daily.
  Arms: Part 2: RO5503781 + Cytarabine; Part 4: Optimized RO5503781 + Cytarabine; Part3:RO5503781+Cytarabine+Anthracycline

SUMMARY:
This Phase 1/1b, open-label study will evaluate the safety and pharmacokinetics of escalating doses of RO5503781 as a single agent or in combination with cytarabine in participants with acute myelogenous leukemia. In Part 1, RO5503781 will be administered in escalating doses as a single agent, and in Part 2, RO5503781 will be administered in combination with cytarabine. An optional Part 3 in which RO5503781 will be administered with cytarabine and anthracycline may be considered . In Part 4, the safety and pharmacokinetic profile of an optimized formulation of RO5503781 in combination with cytarabine will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Documented/confirmed acute myelogenous leukemia (AML), except for acute promyelocytic leukemia
* Eastern Cooperative Oncology Group (ECOG) performance status 0 to 2 in Part 1 and Part 2, participants enrolled in the extension/tail portion, Part 3 and Part 4 must have an ECOG performance status of 0 or 1
* All non-hematological adverse events of any prior chemotherapy, surgery or radiotherapy must have resolved to National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE) Grade less than or equal to (</=) 2 prior to starting therapy
* Adequate hepatic and renal function
* Willing to submit the blood sampling and bone marrow sampling required by protocol

Additional inclusion criteria for Parts 1-4 may apply.

Exclusion Criteria:

* Participants receiving any other investigational or commercial agents or therapies administered with the intention to treat their malignancy within 14 days of first receipt of study drug, with the exception of hydroxyurea as defined in protocol
* History of allergic or toxic reactions attributed to cytarabine (Part 2) or history of allergic reactions to components of the formulated product
* Current evidence of central nervous system (CNS) leukemia
* Participants with severe and/or uncontrolled medical conditions or other conditions that could affect their participation in the study
* Participants with evidence of electrolyte imbalance greater than or equal to (>/=) Grade 2 which cannot be corrected prior to study initiation
* Pregnant or breastfeeding women
* Human immunodeficiency virus (HIV) - positive participants receiving anti-retroviral therapy
* Participants who refuse to potentially receive blood products and/or have a hypersensitivity to blood products

Additional exclusion criteria for Parts 1-4 may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2013-02; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) and/ or Recommended Phase 2 Dose (RP2D) of RO5503781 | Day 1 up to Day 42
Proportion of Participants with Dose-Limiting Toxicities (DLTs) | Day 1 up to Day 42
Safety: Proportion of Participants with Adverse Events (AEs) and Serious Adverse Events (SAEs) | Baseline up to approximately 2 years

SECONDARY OUTCOMES:
Pharmacokinetics: Maximum Observed Plasma Concentration (Cmax) (in Micrograms per Milliliters [mcg/mL]) of RO5503781, Cytarabine,1-beta-D-Arabinofuranosyluracil, Daunorubicin, Daunorubicinol, Idarubicin, and Idarubicinol | Predose (0 Hr) on Cycle (Cy) 1 Day 1 up to Cy 1 Day 15 (Cy length=28 days) (detailed timeframe for individual drug is provided in outcome measure description)
  Timeframe for RO5503781: Predose (0 hour [Hr]), and 1, 2, 3, 4, 6, 10 Hr Postdose on Cy 1 Days 1, 5; Predose (0 Hr) on Cy 1 Day 2; Cy1 Day 6; Cy 1 Days 8, 9, 15 (Parts 1, 2, 4 only) (Cy length=28 days) Timeframe for cytarabine, 1-beta-D-arabinofuranosyluracil (cytarabine metabolite): Parts 2,4: Predose (0Hr), 1, 2, 3, 4, 6, 10 Hr Postdose on Cy1 Days 1, 5; Predose (0Hr) on Cy1 Day 2; Cy1 Day 6; Cy 1 Days 8, 9, 15; Part 3: Predose (0 Hr) on Cy1 Day 1; Predose (0 Hr), 1, 2, 3, 4, 6, 10 Hr Postdose on Cy1 Day 5; Cy1 Day 6 (Cy=28days) Timeframe for daunorubicin, daunorubicinol (daunorubicin metabolite), idarubicin, and idarubicinol (idarubicin metabolite): Part 3: Predose (0 Hr), and 1, 2, 3, 4, 6, 10 Hr Postdose on Cy 1 Days 1, 5; Predose (0 Hr) on Cy1 Day 2; Cy1 Day 6 (Cy length=28 days)
Pharmacokinetics: Time to Reach Maximum Plasma Concentrations (Tmax) in hours of RO5503781, Cytarabine, 1-beta-D-Arabinofuranosyluracil, Daunorubicin, Daunorubicinol, Idarubicin, and Idarubicinol | Predose (0 Hr) on Cy1 Day 1 up to Cy 1 Day 15 (Cy length=28 days) (detailed timeframe for individual drug is provided in outcome measure description).
  Timeframe for RO5503781: Predose (0 hour [Hr]), and 1, 2, 3, 4, 6, 10 Hr Postdose on Cy 1 Days 1, 5; Predose (0 Hr) on Cy 1 Day 2; Cy1 Day 6; Cy 1 Days 8, 9, 15 (Parts 1, 2, 4 only) (Cy length=28 days) Timeframe for cytarabine, 1-beta-D-arabinofuranosyluracil (cytarabine metabolite): Parts 2,4: Predose (0Hr), 1, 2, 3, 4, 6, 10 Hr Postdose on Cy1 Days 1, 5; Predose (0Hr) on Cy1 Day 2; Cy1 Day 6; Cy 1 Days 8, 9, 15; Part 3: Predose (0 Hr) on Cy1 Day 1; Predose (0 Hr), 1, 2, 3, 4, 6, 10 Hr Postdose on Cy1 Day 5; Cy1 Day 6 (Cy=28days) Timeframe for daunorubicin, daunorubicinol (daunorubicin metabolite), idarubicin, and idarubicinol (idarubicin metabolite): Part 3: Predose (0 Hr), and 1, 2, 3, 4, 6, 10 Hr Postdose on Cy 1 Days 1, 5; Predose (0 Hr) on Cy1 Day 2; Cy1 Day 6 (Cy length=28 days)
Pharmacokinetics: Terminal Half-Life (t1/2) (in hours) of RO5503781, Cytarabine, 1-beta-D-Arabinofuranosyluracil, Daunorubicin, Daunorubicinol, Idarubicin, and Idarubicinol | Predose (0 Hr) on Cy1 Day 1 up to Cy 1 Day 15 (Cy length=28 days) (detailed timeframe for individual drug is provided in outcome measure description)
  Timeframe for RO5503781: Predose (0 hour [Hr]), and 1, 2, 3, 4, 6, 10 Hr Postdose on Cy 1 Days 1, 5; Predose (0 Hr) on Cy 1 Day 2; Cy1 Day 6; Cy 1 Days 8, 9, 15 (Parts 1, 2, 4 only) (Cy length=28 days) Timeframe for cytarabine, 1-beta-D-arabinofuranosyluracil (cytarabine metabolite): Parts 2,4: Predose (0Hr), 1, 2, 3, 4, 6, 10 Hr Postdose on Cy1 Days 1, 5; Predose (0Hr) on Cy1 Day 2; Cy1 Day 6; Cy 1 Days 8, 9, 15; Part 3: Predose (0 Hr) on Cy1 Day 1; Predose (0 Hr), 1, 2, 3, 4, 6, 10 Hr Postdose on Cy1 Day 5; Cy1 Day 6 (Cy=28days) Timeframe for daunorubicin, daunorubicinol (daunorubicin metabolite), idarubicin, and idarubicinol (idarubicin metabolite): Part 3: Predose (0 Hr), and 1, 2, 3, 4, 6, 10 Hr Postdose on Cy 1 Days 1, 5; Predose (0 Hr) on Cy1 Day 2; Cy1 Day 6 (Cy length=28 days)
Pharmacokinetics: Area Under Plasma Concentration-Time Curve Over One Dosing Internal (AUCtau) (in mcg*hour/mL) of RO5503781, Cytarabine, 1-beta-D-Arabinofuranosyluracil, Daunorubicin, Daunorubicinol, Idarubicin, and Idarubicinol | Predose (0 Hr) on Cy1 Day 1 up to Cy 1 Day 15 (Cy length=28 days) (detailed timeframe for individual drug is provided in outcome measure description)
  Timeframe for RO5503781: Predose (0 hour [Hr]), and 1, 2, 3, 4, 6, 10 Hr Postdose on Cy 1 Days 1, 5; Predose (0 Hr) on Cy 1 Day 2; Cy1 Day 6; Cy 1 Days 8, 9, 15 (Parts 1, 2, 4 only) (Cy length=28 days) Timeframe for cytarabine, 1-beta-D-arabinofuranosyluracil (cytarabine metabolite): Parts 2,4: Predose (0Hr), 1, 2, 3, 4, 6, 10 Hr Postdose on Cy1 Days 1, 5; Predose (0Hr) on Cy1 Day 2; Cy1 Day 6; Cy 1 Days 8, 9, 15; Part 3: Predose (0 Hr) on Cy1 Day 1; Predose (0 Hr), 1, 2, 3, 4, 6, 10 Hr Postdose on Cy1 Day 5; Cy1 Day 6 (Cy=28days) Timeframe for daunorubicin, daunorubicinol (daunorubicin metabolite), idarubicin, and idarubicinol (idarubicin metabolite): Part 3: Predose (0 Hr), and 1, 2, 3, 4, 6, 10 Hr Postdose on Cy 1 Days 1, 5; Predose (0 Hr) on Cy1 Day 2; Cy1 Day 6 (Cy length=28 days)
Pharmacokinetics: Area Under Plasma Concentration-Time Curve From 0 to the Last Measurable Concentration (AUClast) (in mcg*hour/mL) of RO5503781, Cytarabine, 1-beta-D-Arabinofuranosyluracil, Daunorubicin, Daunorubicinol, Idarubicin, and Idarubicinol | Predose (0 Hr) on Cy1 Day 1 up to Cy 1 Day 15 (Cy length=28 days) (detailed timeframe for individual drug is provided in outcome measure description)
  Timeframe for RO5503781: Predose (0 hour [Hr]), and 1, 2, 3, 4, 6, 10 Hr Postdose on Cy 1 Days 1, 5; Predose (0 Hr) on Cy 1 Day 2; Cy1 Day 6; Cy 1 Days 8, 9, 15 (Parts 1, 2, 4 only) (Cy length=28 days) Timeframe for cytarabine, 1-beta-D-arabinofuranosyluracil (cytarabine metabolite): Parts 2,4: Predose (0Hr), 1, 2, 3, 4, 6, 10 Hr Postdose on Cy1 Days 1, 5; Predose (0Hr) on Cy1 Day 2; Cy1 Day 6; Cy 1 Days 8, 9, 15; Part 3: Predose (0 Hr) on Cy1 Day 1; Predose (0 Hr), 1, 2, 3, 4, 6, 10 Hr Postdose on Cy1 Day 5; Cy1 Day 6 (Cy=28days) Timeframe for daunorubicin, daunorubicinol (daunorubicin metabolite), idarubicin, and idarubicinol (idarubicin metabolite): Part 3: Predose (0 Hr), and 1, 2, 3, 4, 6, 10 Hr Postdose on Cy 1 Days 1, 5; Predose (0 Hr) on Cy1 Day 2; Cy1 Day 6 (Cy length=28 days)
Pharmacokinetics: Area Under Plasma Concentration-Time Curve From 0 to Infinity (AUCinf) (in mcg*hour/mL) of RO5503781, Cytarabine, 1-beta-D-Arabinofuranosyluracil, Daunorubicin, Daunorubicinol, Idarubicin, and Idarubicinol | Predose (0 Hr) on Cy1 Day 1 up to Cy 1 Day 15 (Cy length=28 days) (detailed timeframe for individual drug is provided in outcome measure description)
  Timeframe for RO5503781: Predose (0 hour [Hr]), and 1, 2, 3, 4, 6, 10 Hr Postdose on Cy 1 Days 1, 5; Predose (0 Hr) on Cy 1 Day 2; Cy1 Day 6; Cy 1 Days 8, 9, 15 (Parts 1, 2, 4 only) (Cy length=28 days) Timeframe for cytarabine, 1-beta-D-arabinofuranosyluracil (cytarabine metabolite): Parts 2,4: Predose (0Hr), 1, 2, 3, 4, 6, 10 Hr Postdose on Cy1 Days 1, 5; Predose (0Hr) on Cy1 Day 2; Cy1 Day 6; Cy 1 Days 8, 9, 15; Part 3: Predose (0 Hr) on Cy1 Day 1; Predose (0 Hr), 1, 2, 3, 4, 6, 10 Hr Postdose on Cy1 Day 5; Cy1 Day 6 (Cy=28days) Timeframe for daunorubicin, daunorubicinol (daunorubicin metabolite), idarubicin, and idarubicinol (idarubicin metabolite): Part 3: Predose (0 Hr), and 1, 2, 3, 4, 6, 10 Hr Postdose on Cy 1 Days 1, 5; Predose (0 Hr) on Cy1 Day 2; Cy1 Day 6 (Cy length=28 days)
Pharmacokinetics: Apparent Oral Clearance (CL/F) (in liters/hour) of RO5503781, Cytarabine, 1-beta-D-Arabinofuranosyluracil, Daunorubicin, Daunorubicinol, Idarubicin, and Idarubicinol | Predose (0 Hr) on Cy1 Day 1 up to Cy 1 Day 15 (Cy length=28 days) (detailed timeframe for individual drug is provided in outcome measure description)
  Timeframe for RO5503781: Predose (0 hour [Hr]), and 1, 2, 3, 4, 6, 10 Hr Postdose on Cy 1 Days 1, 5; Predose (0 Hr) on Cy 1 Day 2; Cy1 Day 6; Cy 1 Days 8, 9, 15 (Parts 1, 2, 4 only) (Cy length=28 days) Timeframe for cytarabine, 1-beta-D-arabinofuranosyluracil (cytarabine metabolite): Parts 2,4: Predose (0Hr), 1, 2, 3, 4, 6, 10 Hr Postdose on Cy1 Days 1, 5; Predose (0Hr) on Cy1 Day 2; Cy1 Day 6; Cy 1 Days 8, 9, 15; Part 3: Predose (0 Hr) on Cy1 Day 1; Predose (0 Hr), 1, 2, 3, 4, 6, 10 Hr Postdose on Cy1 Day 5; Cy1 Day 6 (Cy=28days) Timeframe for daunorubicin, daunorubicinol (daunorubicin metabolite), idarubicin, and idarubicinol (idarubicin metabolite): Part 3: Predose (0 Hr), and 1, 2, 3, 4, 6, 10 Hr Postdose on Cy 1 Days 1, 5; Predose (0 Hr) on Cy1 Day 2; Cy1 Day 6 (Cy length=28 days)
Pharmacokinetics: Apparent Volume of Distribution (V/F) (in liters) of RO5503781, Cytarabine, 1-beta-D-Arabinofuranosyluracil, Daunorubicin, Daunorubicinol, Idarubicin, and Idarubicinol | Predose (0 Hr) on Cy 1 Day 1 up to Cy 1 Day 15 (Cy length=28 days) (detailed timeframe for individual drug is provided in outcome measure description)
  Timeframe for RO5503781: Predose (0 hour [Hr]), and 1, 2, 3, 4, 6, 10 Hr Postdose on Cy 1 Days 1, 5; Predose (0 Hr) on Cy 1 Day 2; Cy1 Day 6; Cy 1 Days 8, 9, 15 (Parts 1, 2, 4 only) (Cy length=28 days) Timeframe for cytarabine, 1-beta-D-arabinofuranosyluracil (cytarabine metabolite): Parts 2,4: Predose (0Hr), 1, 2, 3, 4, 6, 10 Hr Postdose on Cy1 Days 1, 5; Predose (0Hr) on Cy1 Day 2; Cy1 Day 6; Cy 1 Days 8, 9, 15; Part 3: Predose (0 Hr) on Cy1 Day 1; Predose (0 Hr), 1, 2, 3, 4, 6, 10 Hr Postdose on Cy1 Day 5; Cy1 Day 6 (Cy=28days) Timeframe for daunorubicin, daunorubicinol (daunorubicin metabolite), idarubicin, and idarubicinol (idarubicin metabolite): Part 3: Predose (0 Hr), and 1, 2, 3, 4, 6, 10 Hr Postdose on Cy 1 Days 1, 5; Predose (0 Hr) on Cy1 Day 2; Cy1 Day 6 (Cy length=28 days)
Pharmacokinetics: Apparent Elimination Rate Constant (kel) (in 1/hour) of RO5503781, Cytarabine, 1-beta-D-Arabinofuranosyluracil, Daunorubicin, Daunorubicinol, Idarubicin, and Idarubicinol | Predose (0 Hr) on Cy 1 Day 1 up to Cy 1 Day 15 (Cy length=28 days) (detailed timeframe for individual drug is provided in outcome measure description)
  Timeframe for RO5503781: Predose (0 hour [Hr]), and 1, 2, 3, 4, 6, 10 Hr Postdose on Cy 1 Days 1, 5; Predose (0 Hr) on Cy 1 Day 2; Cy1 Day 6; Cy 1 Days 8, 9, 15 (Parts 1, 2, 4 only) (Cy length=28 days) Timeframe for cytarabine, 1-beta-D-arabinofuranosyluracil (cytarabine metabolite): Parts 2,4: Predose (0Hr), 1, 2, 3, 4, 6, 10 Hr Postdose on Cy1 Days 1, 5; Predose (0Hr) on Cy1 Day 2; Cy1 Day 6; Cy 1 Days 8, 9, 15; Part 3: Predose (0 Hr) on Cy1 Day 1; Predose (0 Hr), 1, 2, 3, 4, 6, 10 Hr Postdose on Cy1 Day 5; Cy1 Day 6 (Cy=28days) Timeframe for daunorubicin, daunorubicinol (daunorubicin metabolite), idarubicin, and idarubicinol (idarubicin metabolite): Part 3: Predose (0 Hr), and 1, 2, 3, 4, 6, 10 Hr Postdose on Cy 1 Days 1, 5; Predose (0 Hr) on Cy1 Day 2; Cy1 Day 6 (Cy length=28 days)
Pharmacodynamics: Macrophage Inhibitory Cytokine-1 (MIC1) Serum Levels | Predose (0 Hr), and 1, 2, 3, 4, 6, 10 Hr postdose on Cy 1 Days 1, 5; predose (0 Hr) on Cy1 Day 2; Cy1 Day 6; Cy 1 Days 8, 9, 15 (Parts 1, 2, 4 only) (Cy length=28 days)
Pharmacodynamics: Proportion of Participants With Tumor Suppressor Protein 53 (p53) Mutation, as Assessed by Gene Sequencing and/or Research-Use AmpliChip p53 Test | Predose (0 Hr), and 6 Hr postdose on Cy 1 Days 1, 5; predose (0 Hr) on Cy 1 Day 2; Cy 1 Day 6; at disease progression/relapse (up to approximately 3.25 years)
Pharmacodynamics: Murine Double Minute-2 (MDM2) Messenger Ribonucleic Acid (mRNA) Expression, as Assessed by Quantitative Real Time Polymerase Chain Reaction (RT-PCR) | Predose (0 Hr), and 6 Hr postdose on Cy 1 Days 1, 5; predose (0 Hr) on Cy 1 Day 2; Cy 1 Day 6; at disease progression/relapse (up to approximately 3.25 years)
Proportion of Participants With Complete Remission (CR) as best response during study and follow up period, as Assessed Using Bone Marrow and Hematological Examinations | Day 1 of each treatment cycle starting from Cy 2 up to 28 days after last dose of RO5503781 (approximately 3.25 years); additionally, every 2 months for participants with CR from occurrence of CR to 1 year (overall up to approximately 3.25 years)
Proportion of Participants With Complete Remission Without Platelet Recovery (CRp) as best response during study and follow up period as Assessed Using Bone Marrow and Hematological Examinations | Day 1 of each treatment cycle starting from Cy 2 up to 28 days after last dose of RO5503781 (approximately 3.25 years); additionally, every 2 months for participants with CRp from occurrence of CRp to 1 year (overall up to approximately 3.25 years)
Proportion of Participants With Complete Remission With Insufficient Recovery of Peripheral Counts (CRi) or Morphologic Leukemia Free State (MLFS) as Best Response During Study and Follow Up as Assessed Using Bone Marrow and Hematological Examinations | Day 1 of each treatment cycle starting from Cy 2 up to 28 days after last dose of RO5503781 (approximately 3.25 years); additionally, every 2 months for participants with CRi from occurrence of CRi to 1 year (overall up to approximately 3.25 years)
Proportion of Participants With Partial Response (PR) as Best Response During Study and Follow Up Period, as Assessed Using Bone Marrow and Hematological Examinations | Day 1 of each treatment cycle starting from Cy 2 up to 28 days after last dose of RO5503781 (approximately 3.25 years); additionally, every 2 months for participants with PR from occurrence of PR to 1 year (overall up to approximately 3.25 years)
Proportion of Participants With Hematologic Improvement (SD/HI) as Best Response During Study and Follow Up Period, as Assessed Using Bone Marrow and Hematological Examinations | Day 1 of each treatment cycle starting from Cy 2 up to 28 days after last dose of RO5503781 (approximately 3.25 years); additionally, every 2months for participants with SD/HI from occurrence of SD/HI to 1 year (overall up to approximately 3.25years)
Proportion of Participants With Disease Progression as Best Response During Study and Follow Up Period | Baseline up to approximately 3.25 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (12):
- United States (4):
  - USC Norris Cancer Center, Los Angeles, California
  - New York Medical College, Valhalla, New York
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Cancer Therapy & Research Ctr; Dept Institute for Drug Development, San Antonio, Texas
- Peter Maccallum Cancer Centre, Melbourne, Victoria, Australia
- Canada (2):
  - University Health Network; Princess Margaret Hospital; Medical Oncology Dept, Toronto, Ontario
  - McGill University; Sir Mortimer B Davis Jewish General Hospital; Oncology, Montreal, Quebec
- Institut J Paoli I Calmettes; Onco Hematologie 2, Marseille, France
- Azienda Ospedaliera Universitaria Policlinico Sant'Orsola Malpigh, Bologna, Emilia-Romagna, Italy
- South Korea (2):
  - Seoul National Uni Hospital; Dept. of Internal Medicine/Hematology/Oncology, Seoul
  - Asan Medical Center, Seoul
- The Beatson West of Scotland Cancer Centre; Cancer Clinical Trials Unit, Glasgow, United Kingdom

REFERENCES:
- [Derived] Yee K, Papayannidis C, Vey N, Dickinson MJ, Kelly KR, Assouline S, Kasner M, Seiter K, Drummond MW, Yoon SS, Lee JH, Blotner S, Jukofsky L, Pierceall WE, Zhi J, Simon S, Higgins B, Nichols G, Monnet A, Muehlbauer S, Ott M, Chen LC, Martinelli G. Murine double minute 2 inhibition alone or with cytarabine in acute myeloid leukemia: Results from an idasanutlin phase 1/1b study small star, filled. Leuk Res. 2021 Jan;100:106489. doi: 10.1016/j.leukres.2020.106489. Epub 2020 Dec 1. PMID 33302031